CLINICAL TRIAL: NCT03831061
Title: Intervention Through Cognitive Stimulation in People Aged 65 or Older With Mild Cognitive Impairment in Primary Care
Brief Title: Cognitive Stimulation in Older With Mild Cognitive Impairment
Acronym: Cognitive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Isabel Gómez-Soria, Clinical Professor, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: School of Health Sciences
Record Dates: First submitted 2019-01-17; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Mild Cognitive Impairment; Randomized Controlled Trial
Keywords: Mild Cognitive Impairment; Elderly; Randomized Controlled Trial; Cognitive Stimulation; Cognitive Intervention
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: An intervention group and a control group with the same characteristics are included.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cognitive stimulation (Experimental): 10 sessions of 45 minutes/week during 10 weeks. Each session included : (a) temporo-spatial orientation , (b) activities related to memory, orientation, language, praxis, gnosis, calculation, perception, reasoning, visual attention, and executive functions, (c) individual practical exercises and (d) correction of the practical exercises.
  There are 54 participants subdivided into two groups of 27 participants that perform the same intervention in different days of the week.
  Interventions: Other: Cognitive stimulation
- Control group (No intervention) (No Intervention): There are 68 participants in total. These participants did not receive intervention.

INTERVENTIONS:
Other: Cognitive stimulation
  Arms: Cognitive stimulation

SUMMARY:
The participants who carry out our program of cognitive stimulation, deteriorate at a cognitive level more slowly and can improve their score of the Spanish version of 35 points of Mini-mental State of Folstein; Mini-exam Cognoscitive of Lobo.

DETAILED DESCRIPTION:
The aim of our research is to evaluate the effect of a cognitive stimulation program in people aged 65 or older with mild cognitive impairment (MCI) and compare it, in the short, medium and long term, with the evolution of other people, with the same characteristics and for which this intervention has not been carried out.

The significant increase in the number of people over 65 years of age in relation to the total population, suggests a significant increase in age-related pathologies. The problem that entails population aging increases when cognitive deterioration appears.

From an economic perspective, the cognitive deterioration of the elderly person is estimated to contribute to health expenses of almost ten times more compared to people of the same age with cognitive functions preserved. Different studies show that a considerable proportion of people with MCI have a high risk of developing dementia and Alzheimer's disease.

Cognitive stimulation is a treatment that has shown profitability and has been recommended as the treatment of choice in MCI.

Our research is based on a cognitive stimulation that uses the Red Book of Mental Activation. The book consists of 4 practical exercises that work 10 cognitive aspects (memory, orientation, language, praxis, gnosis, calculation, perception, reasoning, attention and programming); in total 40 exercises. The models on which the notebook is based is the cognitive model and the human occupation model.

In the Health Center San José Norte-Centro of Zaragoza (Spain), assessments were made to 416 volunteer candidates, of which 294 were excluded for not meeting the inclusion criteria; being a total of 122 participants that have been part of the randomized controlled trial. Of the 122 participants; 54 have carried out the intervention as an intervention group and 68 as the control group. The control group did not perform any type of intervention.

The intervention was carried out at the La Caridad de Zaragoza Foundation (Spain), consisting of 10 sessions of 45 minutes/week during 10 weeks. The conceptual framework of this intervention is formed by the International Classification of Functioning and Disability (CIF), the framework for practice of Occupational Therapy , the cognitive model and the human occupation model of Gary Kielhofner .

To homogenize both the assessments and the intervention, a standardized training was carried out for the occupational therapists who carried them out and consisted of a theoretical part and a practical part of 10 hours each.

The study began in December 2011, obtained the authorization of the Directorate of Primary Care of the Zaragoza II Sector and the approval of the project by the Research Ethics Committee of the Government of Aragon (CEICA). This study has followed the ethical standards recognized by the Declaration of Helsinki. The initial assessments began this month. The necessary sample size was reached in October 2012 and, from that moment on, randomization and intervention with the selected participants was carried out. Three other assessments were made, both for the intervention group and for the control group, immediately after the intervention, six months and one year after the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Older adults (age ≥ 65)
* Community (not institutionalized)
* Mini-Examen Cognoscitive (MEC) score 24-27 points
* Barthel index > 60 points
* No received cognitive stimulation in the last year
* Hearing problems that interfere with the intervention
* Blindness or vision problems that interfere with the intervention
* Neuropsychiatric disorders (agitation, delusions or hallucinations)
* Motor difficulties that interfere with the intervention.

Exclusion Criteria:

- No agree to participate and no sign the informed consent.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 122 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2012-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The Spanish versions of the Mini-Mental State Examination (MEC-35), | baseline and change in 1 week, 6 months, baseline and 12 moths
  It is a reliable and used instrument for the evaluation of cognitive impairment. It meets criteria of "feasibility", "content validity", "procedural" and "construction". Test-retest reliability: weighted kappa = 0.667, sensitivity = 89.8%, and specificity = 83.9%; with the cutoff point 23/24. A score of 28 is considered the lower limit of normal performance in adult population; scores equal or less than 27 would denote cognitive deficits.

SECONDARY OUTCOMES:
The Barthel Index (Barthel) | baseline and change in 1 week, 6 months, baseline and 12 moths
  Developed by Mahoney & Barthel (1965), assesses the level of independence in ten Basic Activities of Daily Living (BADLs) and is an indicator of skills for people with reduced mobility. Its internal consistency is 0.89-0.92; obtains intra-observer reliability with kappa indexes between 0.47 to 1.0. Values the ability to perform ten BADLs: feeding, bathing, dressing, grooming, bowel control, bladder control, toilet use, transfers chair-bed, mobility and stairs use. A score is assigned to each item (0, 5, 10, 15) as a function of time and help needed. The final score varies from 0 (completely dependent) to 100 (completely independent). Above 60 points there is a high probability of continuing to live in the community.
The scale of Lawton & Brody (Lawton) | baseline and change in 1 week, 6 months, baseline and 12 moths
  Assesses the degree of autonomy in eight Instrumental Activity Daily Livings (IADLs) necessary for living independently in the community. Its reliability is = 0.85 , sensitivity = 0.57 and specificity = 0.92. In a study in Spanish population the internal consistency was 0.94; Regarding the convergent validity all the correlation coefficients were higher than 0.40. A summary score ranges from 0 (low function, dependent) to 8 (high function, independent) for women, and 0 through 5 for men (historically, for men, the areas of food preparation, housekeeping, laundering are excluded).
The Goldberg questionnaire (EADG) | baseline and change in 1 week, 6 months, baseline and 12 moths
  Evaluates the mood referred to anxiety and depresión. The original questionnaire was developed by Goldberg and consisted of 18 items. Consists of two sub-scales, one of anxiety and other of depression. The last 5 questions of the EADG are only formulated if there are positive answers to the first 4 questions, which are obligatory. The higher the number, the more severe your depression is likely to be. Of all the cutoff points, the most suitable result for the sub-scale of anxiety is 4 points and for the sub-scale of depression is 2 point. The Spanish version of EADG has demonstrated its reliability and validity in the field of Primary Care; with a sensitivity of 83.1%, a specificity of 81.8%, a misclassified index of 17.7% and a positive predictive value of 95.3% .
  The investigators used the sub-scale of anxiety; its overall specificity = 91% and its sensitivity = 86%
The abbreviated Yesavage depression scale (GDS-15) | baseline and change in 1 week, 6 months, baseline and 12 moths
  Evaluates the mood referred to depression. The first version consisted of 30 items . Subsequently, abbreviated version (GDS-15) was published with 15 questions; for use in older people living in the community. For cut-off point 4/5 the sensitivity rates vary between 92.7% and 97.0%, the specificity between 54.8% and 65.2%; the positive predictive value between 69.6% and 82.6% and the negative between 83.3% and 94.4%.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldberg DP, Bridges K, Duncan-Jones P, Grayson D. Dimensions of neuroses seen in primary-care settings. Psychol Med. 1987 May;17(2):461-70. doi: 10.1017/s0033291700025022. PMID 3602238
- [Background] Goldberg D, Bridges K, Duncan-Jones P, Grayson D. Detecting anxiety and depression in general medical settings. BMJ. 1988 Oct 8;297(6653):897-9. doi: 10.1136/bmj.297.6653.897. PMID 3140969
- [Background] Lawton MP, Brody EM. Assessment of older people: self-maintaining and instrumental activities of daily living. Gerontologist. 1969 Autumn;9(3):179-86. No abstract available. PMID 5349366
- [Background] Lobo A, Saz P, Marcos G, Dia JL, De-la-Camara C. The prevalence of dementia and depression in the elderly community in a southern European population. The Zaragoza study. Arch Gen Psychiatry. 1995 Jun;52(6):497-506. doi: 10.1001/archpsyc.1995.03950180083011. PMID 7771920
- [Background] Lobo A, Saz P, Marcos G, Dia JL, de la Camara C, Ventura T, Morales Asin F, Fernando Pascual L, Montanes JA, Aznar S. [Revalidation and standardization of the cognition mini-exam (first Spanish version of the Mini-Mental Status Examination) in the general geriatric population]. Med Clin (Barc). 1999 Jun 5;112(20):767-74. Spanish. PMID 10422057
- [Background] Loewen SC, Anderson BA. Reliability of the Modified Motor Assessment Scale and the Barthel Index. Phys Ther. 1988 Jul;68(7):1077-81. doi: 10.1093/ptj/68.7.1077. PMID 3387463
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] Moher D, Schulz KF, Altman D; CONSORT Group. The CONSORT Statement: revised recommendations for improving the quality of reports of parallel-group randomized trials 2001. Explore (NY). 2005 Jan;1(1):40-5. doi: 10.1016/j.explore.2004.11.001. PMID 16791967
- [Background] Monton C, Perez Echeverria MJ, Campos R, Garcia Campayo J, Lobo A. [Anxiety scales and Goldberg's depression: an efficient interview guide for the detection of psychologic distress]. Aten Primaria. 1993 Oct 15;12(6):345-9. Spanish. PMID 8218816
- [Background] Petersen RC. Mild cognitive impairment clinical trials. Nat Rev Drug Discov. 2003 Aug;2(8):646-53. doi: 10.1038/nrd1155. No abstract available. PMID 12904814
- [Background] Petersen RC. Mild Cognitive Impairment. Continuum (Minneap Minn). 2016 Apr;22(2 Dementia):404-18. doi: 10.1212/CON.0000000000000313. PMID 27042901
- [Background] Roley SS, DeLany JV, Barrows CJ, Brownrigg S, Honaker D, Sava DI, Talley V, Voelkerding K, Amini DA, Smith E, Toto P, King S, Lieberman D, Baum MC, Cohen ES, Cleveland PA, Youngstrom MJ; American Occupational Therapy Association Commission on Practice. Occupational therapy practice framework: domain & practice, 2nd edition. Am J Occup Ther. 2008 Nov-Dec;62(6):625-83. doi: 10.5014/ajot.62.6.625. No abstract available. PMID 19024744
- [Background] Shah S, Vanclay F, Cooper B. Improving the sensitivity of the Barthel Index for stroke rehabilitation. J Clin Epidemiol. 1989;42(8):703-9. doi: 10.1016/0895-4356(89)90065-6. PMID 2760661
- [Background] Yesavage JA, Brink TL, Rose TL, Lum O, Huang V, Adey M, Leirer VO. Development and validation of a geriatric depression screening scale: a preliminary report. J Psychiatr Res. 1982-1983;17(1):37-49. doi: 10.1016/0022-3956(82)90033-4. PMID 7183759
- [Result] Arthur A, Jagger C, Lindesay J, Graham C, Clarke M. Using an annual over-75 health check to screen for depression: validation of the short Geriatric Depression Scale (GDS15) within general practice. Int J Geriatr Psychiatry. 1999 Jun;14(6):431-9. PMID 10398352
- [Derived] Gomez-Soria I, Ferreira C, Olivan-Blazquez B, Aguilar-Latorre A, Calatayud E. Effects of cognitive stimulation program on cognition and mood in older adults, stratified by cognitive levels: A randomized controlled trial. Arch Gerontol Geriatr. 2023 Jul;110:104984. doi: 10.1016/j.archger.2023.104984. Epub 2023 Mar 4. PMID 36921506
- [Derived] Gomez-Soria I, Cuenca-Zaldivar JN, Rodriguez-Roca B, Subiron-Valera AB, Salavera C, Marcen-Roman Y, Andrade-Gomez E, Calatayud E. Cognitive Effects of a Cognitive Stimulation Programme on Trained Domains in Older Adults with Subjective Memory Complaints: Randomised Controlled Trial. Int J Environ Res Public Health. 2023 Feb 18;20(4):3636. doi: 10.3390/ijerph20043636. PMID 36834329
- [Derived] Gomez-Soria I, Andres Esteban EM, Gomez Bruton A, Peralta-Marrupe P. [Long-term effect analysis of a cognitive stimulation program in mild cognitive impairment elderly in Primary Care: A randomized controlled trial]. Aten Primaria. 2021 Aug-Sep;53(7):102053. doi: 10.1016/j.aprim.2021.102053. Epub 2021 Apr 14. Spanish. PMID 33865010
- [Derived] Gomez-Soria I, Peralta-Marrupe P, Plo F. Cognitive stimulation program in mild cognitive impairment A randomized controlled trial. Dement Neuropsychol. 2020 Apr-Jun;14(2):110-117. doi: 10.1590/1980-57642020dn14-020003. PMID 32595879